CLINICAL TRIAL: NCT04841577
Title: A Phase 3, Open-label, Randomized, Controlled, Multi-country Study to Evaluate the Immune Response, Safety and Reactogenicity of RSVPreF3 OA Investigational Vaccine When Co-administered With FLU-QIV Vaccine in Adults Aged 60 Years and Above
Brief Title: A Study on the Immune Response and Safety Elicited by a Vaccine Against Respiratory Syncytial Virus (RSV) When Given Alone and Together With a Vaccine Against Influenza in Adults Aged 60 Years and Above
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 214488
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Results first posted 2022-10-18 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Co-Ad Group (Experimental): Participants received 1 dose of RSV_PreF3 Older Adult (OA) investigational vaccine and 1 dose of FLU-QIV at Day 1 and were followed up until the study end.
  Interventions: Biological: RSVPreF3 OA investigational vaccine; Biological: FLU-QIV
- Control Group (Active Comparator): Participants received 1 dose of FLU-QIV at Day 1 and 1 dose of RSV_PreF3 OA investigational vaccine at Day 31 and were followed up until the study end.
  Interventions: Biological: RSVPreF3 OA investigational vaccine; Biological: FLU-QIV

INTERVENTIONS:
Biological: RSVPreF3 OA investigational vaccine — RSVPreF3 OA investigational vaccine administered intramuscularly in the deltoid region of the non-dominant arm.
Biological: FLU-QIV — FLU-QIV administered intramuscularly in the deltoid region of the dominant (Co-Ad Group) arm or the non-dominant (Control Group) arm.

SUMMARY:
The purpose of this study is to assess the immunogenicity, safety and reactogenicity of the RSVPreF3 OA investigational vaccine when co-administered with the seasonal quadrivalent influenza vaccine (FLU-QIV) in adults aged 60 years and above compared to separate administration of the vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Participants, who, in the opinion of the investigator, can and will comply with the requirements of the protocol A male or female ≥60 YOA at the time of the first study intervention administration.
* Participants living in the general community or in an assisted-living facility that provides minimal assistance, such that the participant is primarily responsible for self-care and activities of daily living.
* Written or witnessed informed consent obtained from the participant prior to performance of any study-specific procedure.
* Participants who are medically stable in the opinion of the investigator at the time of first vaccination. Participants with chronic stable medical conditions with or without specific treatment are allowed to participate in this study if considered by the investigator as medically stable.

Exclusion Criteria:

Medical conditions

* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease or immunosuppressive/cytotoxic therapy based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* Hypersensitivity to latex.
* History of GBS, anaphylaxis, febrile seizures, Bell's palsy and narcolepsy.
* Serious or unstable chronic illness.
* Any history of dementia or any medical condition that moderately or severely impairs cognition.
* Recurrent or un-controlled neurological disorders or seizures. Participants with medically-controlled active or chronic neurological diseases can be enrolled in the study as per investigator assessment, provided that their condition will allow them to comply with the requirements of the protocol (e.g. completion of diary cards, attend regular phone calls/study site visits).
* Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.

Prior/Concomitant therapy

* Use of any investigational or non-registered product (drug, vaccine or medical device) other than the study interventions during the period beginning 30 days before the first dose of study vaccines and ending 30 days after the last vaccine administration, or planned use during the study period.
* Administration of an influenza vaccine during the 6 months preceding the study FLU-QIV administration.
* Planned or actual administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first study intervention administration and ending 30 days after the last study intervention administration.

Note: In case an emergency mass vaccination for an unforeseen public health threat is recommended and/or organized by the public health authorities, outside the routine immunization program, the time period described above can be reduced if necessary for that vaccine provided it is used according to the local governmental recommendations and that the Sponsor is notified accordingly.

* Previous vaccination with an RSV vaccine.
* Administration of long-acting immune-modifying drugs or planned administration at any time during the study period).
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 90 days before the first dose of study vaccine or planned administration during the study period.
* Chronic administration (defined as more than 14 consecutive days in total) of immunosuppressants or other immune-modifying drugs during the period starting 90 days prior to the first study vaccination or planned administration during the study period. For corticosteroids, this will mean prednisone ≥20 mg/day, or equivalent. Inhaled and topical steroids are allowed.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug/invasive medical device).

Other exclusions

* History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.
* Planned move during the study conduct that prohibits participation until 1 month post-last vaccine administration.
* Bedridden participants.
* Participation of any study personnel or their immediate dependents, family, or household members.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 976 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2022-02-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- New Zealand (6):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Havelock North
  - GSK Investigational Site, Paraparaumu
  - GSK Investigational Site, Tauranga
  - GSK Investigational Site, Wellington
- GSK Investigational Site, Panama City, Panama
- South Africa (2):
  - GSK Investigational Site, Boksburg, Gauteng
  - GSK Investigational Site, Middelburg, Mpumalanga

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data (IPD) and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Background] Chandler R, Montenegro N, Llorach C, Aguirre LN, Germain S, Kuriyakose SO, Lambert A, Descamps D, Olivier A, Hulstrom V. Immunogenicity, Reactogenicity, and Safety of AS01E-adjuvanted RSV Prefusion F Protein-based Candidate Vaccine (RSVPreF3 OA) When Co-administered With a Seasonal Quadrivalent Influenza Vaccine in Older Adults: Results of a Phase 3, Open-Label, Randomized Controlled Trial. Clin Infect Dis. 2024 Jan 8:ciad786. doi: 10.1093/cid/ciad786. Online ahead of print. PMID 38189778

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 976 participants enrolled in the study, 86 participants were not assigned to any study group and 5 participants did not receive any study treatment.
  885 participants were vaccinated and included in the Exposed Set.
Period: Overall Study
Arm/Group | Co-Ad Group | Control Group
Started | 442 | 443
Completed | 429 | 417
Not Completed | 13 | 26
Not completed — Adverse Event | 5 | 10
Not completed — Lost to Follow-up | 8 | 7
Not completed — CONSENT WITHDRAWAL, NOT DUE TO A (S)AE | 0 | 8
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Co-Ad Group | Control Group | Total
Number analyzed (Participants) | 442 | 443 | 885
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.4 (6.9) | 68.6 (6.9) | 68.5 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 228 | 228 | 456
  Male | 214 | 215 | 429
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 5 | 9
  Black Or African American | 72 | 70 | 142
  Maori | 7 | 5 | 12
  Mixed Race | 218 | 227 | 445
  Native Hawaiian Or Other Pacific Islander | 2 | 1 | 3
  Other, Not Specified | 2 | 0 | 2
  White | 137 | 135 | 272

OUTCOME MEASURES:

1. Primary Outcome: RSV-A Neutralization Antibody Titers Expressed as Geometric Mean Titers (GMTs)
Description: The serum neutralization assay is a functional assay that measures the ability of serum antibodies to neutralize RSV-A entry and replication in a host cell line. The serum neutralizing antibody titer is expressed in ED60 (Estimated Dilution 60) and corresponds to the inverse of the interpolated serum dilution that yields a 60% reduction of the signal compared to a control without serum.
Time Frame: At 1 month after the RSV_PreF3 OA investigational vaccine dose (at Day 31 for the Co-Ad Group and at Day 61 for the Control Group)
Population: The analysis was performed on the Per Protocol set (PPS) which consisted of all eligible participants who received at least 1 study intervention as per protocol, had immunogenicity results pre-post-dose for at least 1 antigen, complied with blood draw intervals and contribution of participants to PPS at specific timepoint will be defined by timepoint, without intercurrent medical conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED 60)
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 427 | 398
Titers (ED 60) | 10060.5 [9126 to 11090.7] | 12255 [11160.4 to 13456.9]
Statistical Analysis 1: Comparison: Co-Ad Group vs Control Group; Adjusted ratios of Control group over Co-Ad Group in RSV-A Neutralizing antibody GMTs at one month after RSV_PreF3 OA investigational vaccination. An Analysis of Covariance (ANCOVA) model was used to analyse post-vaccination log-transformed titers of RSV-A neutralizing antibodies The ANCOVA model included the treatment group, the age category (age at vaccination: 60-69, 70-79 or >=80 years), country and sex as fixed effects and the pre-dose log-10 titer as covariate; Test type: Non-Inferiority — Non-inferiority is demonstrated if the upper limit of the 2-sided 95% confidence interval (CI) of the group GMT ratio [Control group divided by Co Ad group] for RSVPreF3 OA investigational vaccine is ≤ (equal to or smaller than) 1.5; Adjusted group GMT ratio = 1.27, 95% CI 2-sided [1.12 to 1.44]

2. Primary Outcome: Hemagglutinin Inhibition (HI) Antibody Titers for Each of the FLU Vaccine Strains Expressed as Group GMTs
Description: HI antibody titers were assessed for each of the Flu vaccine strains, namely Flu A/Hong Kong/2671/2019 (H3N2), Flu A/Victoria/2570/2019 (H1N1), Flu B/Phuket/3073/2013 (Yamagata) and Flu B/Washington/02/2019 (Victoria). The serum HI antibody titers are expressed in 1/Dilution (DIL) where DIL corresponds to the highest dilution that shows complete HI.
Time Frame: 1 month after the FLU vaccine dose (at Day 31)
Population: The analysis was performed on the PPS which consisted of all eligible participants who received at least 1 study intervention as per protocol, had immunogenicity results pre-post-dose for at least 1 antigen, complied with blood draw intervals and contribution of participants to PPS at specific timepoint will be defined by timepoint, without intercurrent medical conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/DIL)
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 427 | 411
Titers (1/DIL)
  Flu A/Hong Kong/2671/2019 H3N2 | 295.2 [263.6 to 330.6] | 346.8 [306.6 to 392.3]
  Flu A/Victoria/2570/2019 H1N1 | 267.1 [235.6 to 302.8] | 325.4 [282.5 to 374.9]
  Flu B/Phuket/3073/2013 Yamagata | 28.9 [26 to 32.1] | 34.8 [31.1 to 39.0]
  Flu B/Washington/02/2019 Victoria | 41.6 [37.1 to 46.6] | 47.9 [41.9 to 54.8]
Statistical Analysis 1: Comparison: Co-Ad Group vs Control Group; For the Flu A/Hong Kong/2671/2019 (H3N2) strain, an ANCOVA model was used to analyze post-vaccination log-transformed titers. The ANCOVA model included the treatment group, the age category (age at vaccination: 60-69, 70-79 or >=80 years), country and sex as fixed effects and the pre-dose log-10 transformed titer as covariate; Test type: Non-Inferiority — Non-inferiority is demonstrated if the upper limit of the 2-sided 95% confidence interval (CI) of the group GMT ratio [Control group divided by Co Ad group] for each of the FLU vaccine strains is ≤1.5; Adjusted geometric mean titer ratio = 1.17, 95% CI 2-sided [1.02 to 1.35]
Statistical Analysis 2: Comparison: Co-Ad Group vs Control Group; For the Flu A/Victoria/2570/2019 (H1N1) strain, an ANCOVA model was used to analyze post-vaccination log-transformed titers. The ANCOVA model included the treatment group, the age category (age at vaccination: 60-69, 70-79 or >=80 years), country and sex as fixed effects and the pre-dose log-10 transformed titer as covariate; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Adjusted geometric mean Titer ratio = 1.22, 95% CI 2-sided [1.03 to 1.44]
Statistical Analysis 3: Comparison: Co-Ad Group vs Control Group; For the Flu B/Phuket/3073/2013 (Yamagata) strain, an ANCOVA model was used to analyze post-vaccination log-transformed titers. The ANCOVA model included the treatment group, the age category (age at vaccination: 60-69, 70-79 or >=80 years), country and sex as fixed effects and the pre-dose log-10 transformed titer as covariate; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Adjusted geometric mean Titer ratio = 1.17, 95% CI 2-sided [1.04 to 1.32]
Statistical Analysis 4: Comparison: Co-Ad Group vs Control Group; For the Flu B/Washington/02/2019 (Victoria) strain, an ANOVA model was used to analyze post-vaccination log-transformed titers. The ANCOVA model included the treatment group, the age category (age at vaccination: 60-69, 70-79 or >=80 years), country and sex as fixed effects and the pre-dose log-10 transformed titer as covariate; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Adjusted geometric mean Titer ratio = 1.10, 95% CI 2-sided [0.95 to 1.26]

3. Secondary Outcome: Secondary: HI Seroconversion Status for Each of the Flu Vaccine Strains Expressed as Seroconversion Rate (SCR)
Description: SCR for HI antibody response was defined as the percentage of vaccinees who have either a HI pre-dose titer < 1:10 and a post-dose titer >= 1:40 or a pre-dose titer >= 1:10 and at least a four-fold increase in post-dose titer. HI antibody titers were assessed for each of the Flu vaccine strains, namely Flu A/Hong Kong/2671/2019 (H3N2), Flu A/Victoria/2570/2019 (H1N1), Flu B/Phuket/3073/2013 (Yamagata) and Flu B/Washington/02/2019 (Victoria).
Time Frame: 1 month after the FLU vaccine dose (at Day 31)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 427 | 411
Percentage of participants
  Flu A/Hong Kong/2671/2019 H3N2 | 54.3 [49.5 to 59.1] | 56.9 [52.0 to 61.8]
  Flu A/Victoria/2570/2019 H1N1 | 78.9 [74.7 to 82.7] | 83.5 [79.5 to 86.9]
  Flu B/Phuket/3073/2013 Yamagata | 28.8 [24.6 to 33.4] | 32.8 [28.3 to 37.6]
  Flu B/Washington/02/2019 Victoria | 35.6 [31.1 to 40.3] | 36 [31.4 to 40.9]
Statistical Analysis 1: Comparison: Co-Ad Group vs Control Group; For the Flu A/Hong Kong/2671/2019 (H3N2) strain, the 2-sided 95% CI on group difference in seroconversion rate (Control group minus Co-Ad group); Test type: Non-Inferiority — Non-inferiority is demonstrated if the upper limit of the 2-sided 95% CI on the group difference (Control group minus Co-Ad group) in seroconversion rate is ≤10% for HI antibody titers; Miettinen and Nurminen; Difference in percentage = 2.60, 95% CI 2-sided [-4.13 to 9.30]
Statistical Analysis 2: Comparison: Co-Ad Group vs Control Group; For the Flu A/Victoria/2570/2019 (H1N1) strain, the 2-sided 95% CI on group difference in seroconversion rate (Control group minus Co-Ad group); Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Miettinen and Nurminen; Difference in percentage = 4.53, 95% CI 2-sided [-0.77 to 9.83]
Statistical Analysis 3: Comparison: Co-Ad Group vs Control Group; For the Flu B/Phuket/3073/2013 (Yamagata) strain, the 2-sided 95% CI on group difference in seroconversion rate (Control group minus Co-Ad group); Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Miettinen and Nurminen; Difference in percentage = 4.04, 95% CI 2-sided [-2.21 to 10.28]
Statistical Analysis 4: Comparison: Co-Ad Group vs Control Group; For the Flu B/Washington/02/2019 (Victoria) strain, the 2-sided 95% CI on group difference in seroconversion rate (Control group minus Co-Ad group); Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Miettinen and Nurminen; Difference in percentage = 0.41, 95% CI 2-sided [-6.07 to 6.90]

4. Secondary Outcome: RSV-A Neutralization Antibody Titers Expressed as Mean Geometric Increase (MGI)
Description: MGI was defined as the geometric mean of the within participant ratios of the post dose titer over the pre-dose titer.
Time Frame: 1 month after the RSV_PreF3 OA investigational vaccine dose (at Day 31 for the Co-Ad Group and at Day 61 for the Control Group)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 427 | 398
Ratio | 9.61 [8.7 to 10.61] | 12.95 [11.75 to 14.28]

5. Secondary Outcome: RSV-B Neutralization Antibody Titers Expressed as Geometric Mean Titers (GMT)
Description: The serum neutralization assay is a functional assay that measures the ability of serum antibodies to neutralize RSV-B entry and replication in a host cell line. The serum neutralizing antibody titer is expressed in ED60 (Estimated Dilution 60) and corresponds to the inverse of the interpolated serum dilution that yields a 60% reduction of the signal compared to a control without serum.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED 60)
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 212 | 206
Titers (ED 60) | 10518.6 [9302 to 11894.3] | 14349.7 [12640.6 to 16289.9]
Statistical Analysis 1: Comparison: Co-Ad Group vs Control Group; Adjusted ratios of Control group over Co-Ad Group in RSV-B Neutralizing antibody GMTs at one month after RSV_PreF3 OA investigational vaccination. An Analysis of Covariance (ANCOVA) model was used to analyse post-vaccination log-transformed titers of RSV-B neutralizing antibodies. The ANCOVA model included the treatment group, the age category (age at vaccination: 60-69, 70-79 or >=80 years), country and sex as fixed effects and the pre-dose log-10 titer as covariate; Test type: Other; Adjusted group GMT ratio = 1.28, 95% CI 2-sided [1.09 to 1.51]

6. Secondary Outcome: RSV-B Neutralization Antibody Titers Expressed as MGI
Description: MGI was defined as the geometric mean of the within participant ratios of the post-dose titer over the pre-dose titer.
Time Frame: as for outcome 4
Population: The analysis was performed on a subset of the PPS which consisted of all eligible participants who received at least 1 study intervention as per protocol, had immunogenicity results pre-post-dose for at least 1 antigen, complied with blood draw intervals and contribution of participants to PPS at specific timepoint will be defined by timepoint, without intercurrent medical conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 212 | 206
Ratio | 7.67 [6.76 to 8.72] | 9.28 [8.06 to 10.69]

7. Secondary Outcome: HI Antibody Titers for Each of the FLU Vaccine Strains Expressed as GMTs
Description: HI antibody titers were assessed for each of the Flu vaccine strains, namely A/Hong Kong/2671/2019 (H3N2), Flu A/Victoria/2570/2019 (H1N1), Flu B/Phuket/3073/2013 (Yamagata) and Flu B/Washington/02/2019 (Victoria). The serum HI antibody titers are expressed in 1/DIL where DIL corresponds to the highest dilution that shows complete HI.
Time Frame: At baseline (at Day 1) and 1 month after the FLU vaccine dose (at Day 31)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/DIL)
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 435 | 437
Titers (1/DIL)
  Flu A/Hong Kong/2671/2019 H3N2, Day 1 | 61.4 [53.8 to 69.9] | 63.3 [55.7 to 71.9]
  Flu A/Hong Kong/2671/2019 H3N2, Day 31: number analyzed (Participants) | 427 | 411
  Flu A/Hong Kong/2671/2019 H3N2, Day 31 | 295.2 [263.6 to 330.6] | 346.8 [306.6 to 392.3]
  Flu A/Victoria/2570/2019 H1N1, Day 1 | 20 [18 to 22.3] | 19.9 [17.8 to 22.2]
  Flu A/Victoria/2570/2019 H1N1, Day 31: number analyzed (Participants) | 427 | 411
  Flu A/Victoria/2570/2019 H1N1, Day 31 | 267.1 [235.6 to 302.8] | 325.4 [282.5 to 374.9]
  Flu B/Phuket/3073/2013 Yamagata, Day 1 | 10.4 [9.5 to 11.3] | 10.8 [9.9 to 11.7]
  Flu B/Phuket/3073/2013 Yamagata, Day 31: number analyzed (Participants) | 427 | 411
  Flu B/Phuket/3073/2013 Yamagata, Day 31 | 28.9 [26 to 32.1] | 34.8 [31.1 to 39]
  Flu B/Washington/02/2019 Victoria, Day 1 | 12.2 [11.1 to 13.4] | 13.5 [12.2 to 15.1]
  Flu B/Washington/02/2019 Victoria, Day 31: number analyzed (Participants) | 427 | 411
  Flu B/Washington/02/2019 Victoria, Day 31 | 41.6 [37.1 to 46.6] | 47.9 [41.9 to 54.8]

8. Secondary Outcome: HI Seroprotection Status for Each of the FLU Vaccine Strains Expressed as Seroprotection Rate (SPR)
Description: SPR for HI antibody response was defined as percentage of vaccinees with a serum HI titer >= 1:40 that usually is accepted as indicating protection. HI antibody titers were assessed for each of the Flu vaccine strains, namely A/Hong Kong/2671/2019 (H3N2), Flu A/Victoria/2570/2019 (H1N1), Flu B/Phuket/3073/2013 (Yamagata) and Flu B/Washington/02/2019 (Victoria).
Time Frame: At baseline (at Day 1) and 1 month after the FLU vaccine dose (at Day 31)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 435 | 437
Percentage of participants
  Flu A/Hong Kong/2671/2019 H3N2, Day 1 | 70.8 [66.3 to 75] | 70.3 [65.7 to 74.5]
  Flu A/Hong Kong/2671/2019 H3N2, Day 31: number analyzed (Participants) | 427 | 411
  Flu A/Hong Kong/2671/2019 H3N2, Day 31 | 97.4 [95.4 to 98.7] | 97.1 [95 to 98.5]
  Flu A/Victoria/2570/2019 H1N1, Day 1 | 35.4 [30.9 to 40.1] | 34.6 [30.1 to 39.2]
  Flu A/Victoria/2570/2019 H1N1, Day 31: number analyzed (Participants) | 427 | 411
  Flu A/Victoria/2570/2019 H1N1, Day 31 | 94.6 [92 to 96.6] | 93.4 [90.6 to 95.6]
  Flu B/Phuket/3073/2013 Yamagata, Day 1 | 14.3 [11.1 to 17.9] | 14.9 [11.7 to 18.6]
  Flu B/Phuket/3073/2013 Yamagata, Day 31: number analyzed (Participants) | 427 | 411
  Flu B/Phuket/3073/2013 Yamagata, Day 31 | 47.8 [43 to 52.6] | 54.3 [49.3 to 59.2]
  Flu B/Washington/02/2019 Victoria, Day 1 | 20 [16.3 to 24.1] | 23.6 [19.7 to 27.8]
  Flu B/Washington/02/2019 Victoria, Day 31: number analyzed (Participants) | 427 | 411
  Flu B/Washington/02/2019 Victoria, Day 31 | 59.3 [54.4 to 64] | 61.3 [56.4 to 66]

9. Secondary Outcome: HI Antibody Titers for Each of the FLU Vaccine Strains Expressed as MGI
Description: MGI was defined as the geometric mean of the within participant ratios of the post-dose titer over the pre-dose titer. HI antibody were assessed for each of the FLUvaccine strain, namely A/Hong Kong/2671/2019 (H3N2), Flu A/Victoria/2570/2019 (H1N1), Flu B/Phuket/3073/2013 (Yamagata) and Flu B/Washington/02/2019 (Victoria).
Time Frame: 1 month after the FLU vaccine dose (at Day 31)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 427 | 410
Ratio
  Flu A/Hong Kong/2671/2019 H3N2 | 4.81 [4.22 to 5.48] | 5.50 [4.81 to 6.29]
  Flu A/Victoria/2570/2019 H1N1 | 13.36 [11.58 to 15.42] | 16.25 [14.08 to 18.76]
  Flu B/Phuket/3073/2013 Yamagata HI | 2.82 [2.55 to 3.12] | 3.22 [2.90 to 3.58]
  Flu B/Washington/02/2019 Victoria | 3.43 [3.06 to 3.85] | 3.60 [3.18 to 4.08]

10. Secondary Outcome: Percentage of Participants With Solicited Administration Site Events
Description: Solicited administration site adverse events(AEs) assessed were erythema, pain and swelling. Any = occurrence of the adverse event regardless of intensity grade.
Time Frame: Within 4 days (the day of vaccination and 3 subsequent days) after each vaccination
Population: The analysis was performed on the Exposed set, which included All participants who received a study intervention. Analysis per group is based on the study intervention administered. RSV vaccine was administered at day 1 for the control group and at day 31 for the Co-Ad group.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 438 | 438
Percentage of participants
  Erythema against Flu Dose given at Day 1 | 1.1 [0.4 to 2.6] | 0.5 [0.1 to 1.6]
  Erythema against RSV Dose given at Day 1: number analyzed (Participants) | 438 | 0
  Erythema against RSV Dose given at Day 1 | 4.1 [2.5 to 6.4] |
  Erythema against RSV Dose given at Day 31: number analyzed (Participants) | 0 | 419
  Erythema against RSV Dose given at Day 31 |  | 2.1 [1 to 4]
  Pain against Flu Dose given at Day 1 | 28.3 [24.1 to 32.8] | 20.5 [16.9 to 24.6]
  Pain against RSV Dose given at Day 1: number analyzed (Participants) | 438 | 0
  Pain against RSV Dose given at Day 1 | 47.9 [43.2 to 52.7] |
  Pain against RSV Dose give at Day 31: number analyzed (Participants) | 0 | 419
  Pain against RSV Dose give at Day 31 |  | 39.1 [34.4 to 44]
  Swelling against Flu Dose given at Day 1 | 1.4 [0.5 to 3] | 0.7 [0.1 to 2]
  Swelling against RSV Dose given at Day 1: number analyzed (Participants) | 438 | 0
  Swelling against RSV Dose given at Day 1 | 3.2 [1.8 to 5.3] |
  Swelling against RSV Dose given at Day 31: number analyzed (Participants) | 0 | 419
  Swelling against RSV Dose given at Day 31 |  | 1 [0.3 to 2.4]

11. Secondary Outcome: Percentage of Participants With Solicited Systemic Events
Description: Solicited systemic events assessed were arthralgia, fatigue, fever [defined as temperature equal to or above (>=) 38 degrees Celsius (C)/100.4 degrees Fahrenheit (F)], headache and myalgia. Any = occurrence of the adverse event regardless of intensity grade or relation to study vaccination.
Time Frame: Within 4 days (the day of vaccination and 3 subsequent days) after each vaccination
Population: The analysis was performed on the Exposed set, which included All participants who received a study intervention. Analysis per group is based on the study intervention administered. The Co-Ad group only received vaccination at Day 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 438 | 438
Percentage of participants
  Arthralgia, Dosing at Day 1 | 16.2 [12.9 to 20] | 4.8 [3 to 7.2]
  Arthralgia, Dosing at Day 31: number analyzed (Participants) | 0 | 419
  Arthralgia, Dosing at Day 31 |  | 11.2 [8.4 to 14.6]
  Fatigue, Dosing at Day 1 | 22.4 [18.6 to 26.6] | 12.8 [9.8 to 16.3]
  Fatigue, Dosing at Day 31: number analyzed (Participants) | 0 | 419
  Fatigue, Dosing at Day 31 |  | 17.9 [14.3 to 21.9]
  Fever, Dosing at Day 1 | 2.5 [1.3 to 4.4] | 0.7 [0.1 to 2]
  Fever, Dosing at Day 31: number analyzed (Participants) | 0 | 419
  Fever, Dosing at Day 31 |  | 1 [0.3 to 2.4]
  Headache, Dosing at Day 1 | 21.7 [17.9 to 25.8] | 12.8 [9.8 to 16.3]
  Headache, Dosing at Day 31: number analyzed (Participants) | 0 | 419
  Headache, Dosing at Day 31 |  | 16.2 [12.8 to 20.1]
  Myalgia, Dosing at Day 1 | 22.1 [18.3 to 26.3] | 9.4 [6.8 to 12.5]
  Myalgia, Dosing at Day 31: number analyzed (Participants) | 0 | 419
  Myalgia, Dosing at Day 31 |  | 19.6 [15.9 to 23.7]

12. Secondary Outcome: Percentage of Participants Reporting at Least One Unsolicited Adverse Event
Description: An unsolicited AEs is any AE reported in addition to those solicited during the clinical study and that was not included in a list of solicited events using a Participant Diary. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is reported as an unsolicited adverse event. Unsolicited AEs include serious, non-serious AEs and potential immune-mediated diseases (pIMDs). Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within 30 days (the day of vaccination and 29 subsequent days) after each vaccination
Population: The analysis was performed on the Exposed set, which included All participants who received a study intervention. Analysis per group is based on the study intervention administered.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 442 | 443
Percentage of participants | 18.8 [15.2 to 22.7] | 23.7 [19.8 to 27.9]

13. Secondary Outcome: Percentage of Participants Reporting at Least One Serious Adverse Event (SAE)
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant. Any = occurrence of the symptom regardless of intensity grade or relationship to vaccination.
Time Frame: From Day 1 up to study end (6 months after last vaccination)
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 442 | 443
Percentage of Participants | 3.4 [1.9 to 5.5] | 4.5 [2.8 to 6.9]

14. Secondary Outcome: Percentage of Participants Reporting at Least One Potential Immune-mediated Disease (pIMD)
Description: pIMDs are a subset of AEs of special interest that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
Time Frame: From Day 1 up to study end (6 months after last vaccination)
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 442 | 443
Percentage of participants | 1.1 [0.4 to 2.6] | 0.2 [0 to 1.3]

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected during the 4-day follow-up period after vaccination. Unsolicited AEs were collected during the 30-day follow-up period after vaccination. SAEs and pIMDs were collected throughout the study period (from Day 1 to Study end (6 months after last vaccination)).
Arm/Group | Co-Ad Group | Control Group
All-Cause Mortality (participants affected / at risk) | 4/442 | 8/443
Serious Adverse Events (participants affected / at risk) | 15/442 | 20/443
Other Adverse Events (participants affected / at risk) | 290/442 | 276/443
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-Ad Group (N=442) | Control Group (N=443)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 4 (4) | 8 (8)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 3 (3)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Acute disseminated encephalomyelitis (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-Ad Group (N=442) | Control Group (N=443)
Injection site pain (General disorders) | 236 (236) | 192 (254)
Fatigue (General disorders) | 100 (102) | 106 (133)
Injection site erythema (General disorders) | 21 (21) | 11 (11)
Injection site swelling (General disorders) | 16 (16) | 8 (8)
Pyrexia (General disorders) | 14 (14) | 6 (7)
Injection site bruising (General disorders) | 3 (3) | 1 (1)
Injection site pruritus (General disorders) | 1 (1) | 3 (3)
Pain (General disorders) | 3 (3) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 2 (2)
Administration site swelling (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (1)
Injection site discolouration (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 1 (1)
Vaccination site bruising (General disorders) | 0 (0) | 1 (1)
Vaccination site pain (General disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 98 (101) | 100 (125)
Arthralgia (Musculoskeletal and connective tissue disorders) | 73 (73) | 60 (73)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 99 (112) | 103 (134)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 2 (2)
Hypokinesia (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 10 (11)
COVID-19 (Infections and infestations) | 0 (0) | 5 (5)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Tooth abscess (Infections and infestations) | 1 (1) | 2 (2)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Nail infection (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinonasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (3)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 8 (8)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Faecal volume increased (Investigations) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-11-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT04841577/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/77/NCT04841577/SAP_001.pdf